CLINICAL TRIAL: NCT06964867
Title: Effectiveness of Multimedia Health Education to Reduce Anxiety in Patients With Vitreous Floaters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changzhou No.2 People's Hospital (Other)
Responsible Party: Principal Investigator, Qing Feng, Principal Investigator, Changzhou No.2 People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 213001
Record Dates: First submitted 2025-04-22; First posted 2025-05-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Vitreous Floaters; Anxiety
Keywords: vitreous floaters; anxiety; health education; STAI; VFQ-25
MeSH Terms: conditions — vitreous floaters; Anxiety Disorders; Health Education

STUDY DESIGN:
Intervention Model Description: Multimedia health education was designed as an intervention. This intervention was administered by a single vitreoretinal specialist with over a decade of clinical experience. This standardized protocol comprised a 30-minute didactic session utilizing power point presentations (PPT), systematically covering: 1) Etiopathogenesis; 2) Symptomatology; 3) Therapeutic modalities; 4) Follow-up necessity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- the multimedia health education group (Experimental): Multimedia health education was designed as an intervention. This intervention was administered by a single vitreoretinal specialist with over a decade of clinical experience. This standardized protocol comprised a 30-minute didactic session utilizing power point presentations (PPT), systematically covering: 1) Etiopathogenesis: Molecular mechanisms of vitreous syneresis and collagen aggregation; 2) Symptomatology: Characteristic visual phenomena and differential diagnosis; 3) Therapeutic modalities: Evidence hierarchy from observation to vitrectomy (including Nd:YAG laser efficacy controversies); 4) Follow-up necessity: Red flag symptoms warranting urgent re-evaluation (sudden floaters with photopsia)
  Interventions: Other: Multimedia Health Education

INTERVENTIONS:
Other: Multimedia Health Education — Multimedia health education was designed as an intervention. This intervention was administered by a single vitreoretinal specialist with over a decade of clinical experience. This standardized protocol comprised a 30-minute didactic session utilizing power point presentations (PPT), systematically covering: 1) Etiopathogenesis: Molecular mechanisms of vitreous syneresis and collagen aggregation; 2) Symptomatology: Characteristic visual phenomena and differential diagnosis; 3) Therapeutic modalities: Evidence hierarchy from observation to vitrectomy (including Nd:YAG laser efficacy controversies); 4) Follow-up necessity: Red flag symptoms warranting urgent re-evaluation (sudden floaters with photopsia)

SUMMARY:
The patients with vitreous floaters were randomly divided into to groups after excluding the possibility of coexisting ocular pathologies potentially confounding visual symptoms or vitreoretinal anatomy. The control group performed conventional oral education. The experimental group conducted multimedia health education activities on the basis of conventional oral education. Their VRQoL (Visual Function Questionnaire-25, VFQ-25) and anxiety status (State-Trait Anxiety Inventory, STAI) were evaluated before education and at the final follow-up. The demographic and clinical characteristics (gender, age, eduaction, duration of vitreous floaters, comorbidities and so on) were collected.

DETAILED DESCRIPTION:
Patients inclusion criteria: 1)Patients with VF visited the Department of Ophthalmology, the third affiliated hospital of Nanjing Medical University between December 2023 and April 2025; 2) Endogenously derived subjective floaters confirmed by comprehensive ophthalmic examination including slit-lamp biomicroscopy, dilated fundoscopy, optical coherence tomography (OCT) and so on; 3) Willing to participate in the multimedia health education program and complete validated questionnaires, with written informed consent obtained.

exclusion criteria:

1)Secondary VF requiring surgical intervention (e.g., vitreous hemorrhage, retinal breaks, or uveitis); 2) Coexisting ocular pathologies potentially confounding visual symptoms or vitreoretinal anatomy (e.g., diabetic retinopathy, retinal vascular occlusion, epiretinal membrane, or vitreomacular traction syndrome); 3) History of vitreoretinal surgery (PPV or laser procedures); 4) Refusal or inability to complete study protocols.

Intervention:

Multimedia health education was designed as an intervention. This intervention was administered by a single vitreoretinal specialist with over a decade of clinical experience. This standardized protocol comprised a 30-minute didactic session utilizing power point presentations (PPT), systematically covering: 1) Etiopathogenesis: molecular mechanisms of vitreous syneresis and collagen aggregation; 2) Symptomatology: characteristic visual phenomena and differential diagnosis; 3) Therapeutic modalities: evidence hierarchy from observation to vitrectomy (including Nd:YAG laser efficacy controversies); 4) Follow-up necessity: red flag symptoms warranting urgent re-evaluation (sudden floaters with photopsia). Multimedia presentation was made through pictures, texts, sounds, and videos. The simple and easy-to-understand language were used to make population easy to accept.

All participants underwent comprehensive ophthalmic evaluations comprising best-corrected visual acuity (BCVA), slit-lamp biomicroscopy with anterior segment analysis, dilated fundus examination incorporating scanning laser ophthalmoscopy (SLO) and spectral-domain optical coherence tomography (SD-OCT) to exclude vitreoretinal interface pathologies such as epiretinal membranes, macular holes and so on. Demographic and clinical baseline characteristics were systematically recorded, including gender, age, educational attainment, sympotom duration, presence or absence of photopsia, time of using electronic products daily, comorbidities, shape of floaters, diopter, psychometric and visual-related quality of life (VRQoL) assessments using National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) and State-Trait Anxiety Inventory (STAI). To minimize intervention selection bias, a pragmatic temporal allocation protocol was implemented: Patients attending the clinic during odd-numbered calendar weeks were prospectively allocated to the multimedia health education group whereas those presenting during even-numbered weeks comprised the routine verbal group.

At the 3-month follow-up, both groups completed validated the VFQ-25 and STAI-state questionnaires via phone or wechat.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of vitreous floaters;
2. Be able to complete questionnaires.

Exclusion Criteria:

1. Secondary VF requiring surgical intervention;
2. Coexisting ocular pathologies potentially confounding vitreoretinal anatomy;
3. History of vitreoretinal surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory scores | before the intervention, 3months after the intervention
  This questionnaire comprise two 20-item subscales state anxity and trait anxiety: STAI-state evaluating transient emotional responses ("how you feel right now") and STAI-trait measuring stable anxiety predisposition ("how you generally feel"). The scores for each test ranged from 20 to 80 points, with higher scores indicating higher anxiety.Scoring followed Spielberger's manualized criteria. According to the Spielberger manual, STAI-state and STAI-trait are categorized as follows: mild anxiety ranges from 20 to 39, moderate anxiety from 40 to 59, and high anxiety from 60 to 80.

SECONDARY OUTCOMES:
Visual Function Quality 25 scores. | before the intervention, 3months after the intervention
  The scale consists of 12 dimensions empassing 26 items, including one overall health scale and 11 visual related scales. 26 items all scored ranged from 0 to 100 points, The 26 items are scored on a scale from 0 to 100 points. If the patient responds with 1, 2, 3, 4, or 5, the scores are assigned as 0, 25, 50, 75, and 100 points, respectively. A higher scale score indicates better VRQoL, while a lower score reflects poorer visual-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second People's Hospital of Changzhou, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided